CLINICAL TRIAL: NCT05778825
Title: A Pilot Study of Oral Minoxidil for the Treatment of Persistent Hair Loss in Pediatric, Adolescent, and Young Adult Cancer Survivors
Brief Title: A Study of Oral Minoxidil to Treat Hair Loss in Children, Teens, and Young Adults Who Are Cancer Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-022
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Survivors of Childhood Cancer; Alopecia
Keywords: Hair loss; Minoxidil; 23-022
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Minoxidil (Experimental): Patients receive oral minoxidil at a dose of 0.01 (<40kg) and 0.02 (≥40kg) mg/kg/day for 8 months
  Interventions: Drug: Oral Minoxidil
- Placebo followed by oral Minoxidil (Active Comparator): Patient receive placebo for 4 months followed by oral minoxidil for 4 months
  Interventions: Drug: Oral Minoxidil; Other: Placebo

INTERVENTIONS:
Drug: Oral Minoxidil — minoxidil at a dose of 0.01 (<40kg) and 0.02 (≥40kg) mg/kg/day
Other: Placebo — placebo for 4 months
  Arms: Placebo followed by oral Minoxidil

SUMMARY:
This study will test whether minoxidil taken by mouth (oral minoxidil) can improve hair loss caused by cancer treatment in children and young adults. In addition, the researchers will test the safety of oral minoxidil, and see if the study drug causes few or mild side effects in participants. Other purposes of this study include looking at whether participants are able to follow their study drug dosing schedules, and how oral minoxidil affects participants' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been diagnosed with cancer before the age of 17.
* They must have completed either systemic or radiation therapy (cytotoxic chemotherapy and external beam radiation therapy) for their cancer at least 1 year prior to study entry.
* They must be between 6-18 years old at the time of enrollment.
* They must have a clinical diagnosis of persistent or late alopecia for >6 months and that is definitely, probably, or possibly related to prior chemotherapy and/or radiation.

Exclusion Criteria:

* Had a history of alopecia prior to systemic or radiation therapy for cancer, or has alopecia unrelated to cancer treatment.
* Have scalp disorders that preclude the evaluation of alopecia, such as psoriasis
* Has a known hypersensitivity to minoxidil
* Concurrent use of other therapies for alopecia
* Concurrent active anticancer therapies (cytotoxic, targeted, endocrine, immunologic)
* History of chronic sclerotic cutaneous GvHD affecting the scalp
* Active chronic cutaneous GvHD
* History of orthostatic or symptomatic hypotension, syncope related to hypotension; systolic less than or equal than 100 (for adults) and 90 (for children) at screening.
* Pregnancy.
* Cardiovascular disease that in the opinion of the cardiologist makes the patient unsuitable for therapy
* Blood pressure less than the 5th percentile or less than 90/50 mmHg for children 10 years or older

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
change in the target area (1/3 of the distance midline from glabella to occiput from the front toward the back) hair density | at 4 months
  as assessed by Hairmetrix allows trichoscopy (dermoscopic imaging of the scalp and hair) in real time. It requires no special scalp or hair preparation and allows fully automated unclipped analysis, producing measurements.
change in the target area (1/3 of the distance midline from glabella to occiput from the front toward the back) hair density | at 8 months
  as assessed by Hairmetrix allows trichoscopy (dermoscopic imaging of the scalp and hair) in real time. It requires no special scalp or hair preparation and allows fully automated unclipped analysis, producing measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Markova, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm